CLINICAL TRIAL: NCT00732147
Title: Effects of Pramlintide on Endogenous Production of VLDL-Triglyceride and Glucose in the Post Prandial State in Type 2 Diabetes Mellitus
Brief Title: Effects of Pramlintide on Endogenous Production of Very-low-density-lipoprotein (VLDL)-Triglyceride and Glucose in the Post Prandial State in T2DM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor could not fund.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Chair, Department of Medicine; Director, General Clinical Research Center; Director, Clinical and Translational Sciences Institute, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: hp-00044094
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes
Keywords: triglycerides; endogenous; glucose; production
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — pramlintide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Type 2 diabetes patients will receive placebo with 3 meals in experimental period.
  Interventions: Drug: Placebo
- 1 (Experimental): Type 2 Diabetes patient will receive Pramlintide with 3 meals in experimental period.
  Interventions: Drug: Pramlintide acetate

INTERVENTIONS:
Drug: Pramlintide acetate — 120 micrograms given subcutaneously before each meal X 3.
  Other Names: Symlin
  Arms: 1
Drug: Placebo — 120 micrograms given subcutaneously before each meal x 3.
  Arms: 2

SUMMARY:
Diabetes affects almost 21 million people in the United States. In this study we will test a drug called Pramlintide(Symlin), and see how it works to lower blood sugar and fat levels after a meal. Lowering high sugar levels and fat levels after a meal is very important in the prevention of the problems that persons with type 2 diabetes often encounter. Hypothesis is that Pramlintide will lower blood sugar and fat levels after a meal.

DETAILED DESCRIPTION:
A well recognized and troublesome feature of diabetes management is the exacerbated post prandial glucose elevations following a typical high fat meal. To date the mechanisms driving this increased post prandial glycemia are unclear. Pramlintide is believed to affect intermediary metabolism as well as nutrient absorption. The relative contributions from altered absorption and metabolism to the observed post prandial reductions in plasma glucose and TG concentrations remain uncertain, however. Combinations of radioactive and stable isotope labeling techniques are able to quantify the relevant fluxes of glucose and lipids in vivo in humans and are therefore able to provide quantitative answers to these questions.

Aims:

1. To determine the effects of Pramlintide on reducing endogenous production of very-low-density-lipoprotein (VLDL)-triglycerides(TG) following a high fat breakfast, lunch and dinner in patients with type 2 diabetes mellitus (T2DM). A triple isotope approach will be used to determine rate of appearance of (VLDL)-triglycerides following breakfast, lunch and dinner.
2. To compare the relative roles of slowed glucose absorption and reduced endogenous glucose production (glucagonstatic mechanism) in the glucose-lowering effects of Pramlintide in the post prandial state in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM study participants will be C-Peptide positive (levels > 0.3 nmol/L)
* Receiving insulin, metformin and/or sulfonylurea/glitinide.
* Maintained on stable anti-hypertensive medication.
* BMI < 52 kg/m2.
* T2DM for at least 3 months with HBA1C under 10%.

Exclusion Criteria:

* Receiving TZDs, exenatide, sitagliptin or pramlintide therapy.
* Receiving medications known to impair gastric emptying, intestinal motility, glucagon release or corticosteroids.
* Triglyceride levels > 400 mg/dl.
* BMI > 52 kg/m2.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Endogenous glucose production | 18 hours

SECONDARY OUTCOMES:
Endogenous VLDL-Triglyceride production | 18 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — Vanderbilt University